CLINICAL TRIAL: NCT00701168
Title: A Humanitarian Device Exemption Use Protocol of Therasphere® for Treatment of Unresectable Hepatocellular and Metastatic Liver Tumors - HDE #980006
Brief Title: Therasphere® for Treatment of Unresectable Primary Liver Cancer and Metastatic Liver Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Leo W. Jenkins Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LJCC 07-04
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Carcinoma, Hepatocellular; Neoplasm Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis

INTERVENTIONS:
Device: yttrium Y 90 microspheres (Therasphere®) — This is a local therapy for unresectable liver tumors with limited treatment options. It may be repeated under special circumstances.

SUMMARY:
The purpose of this protocol is to provide supervised and limited access to Therasphere® treatment for patients with primary liver cancer and chemotherapy refractory liver metastasis who cannot be treated by surgical removal of the affected part of the liver. Patient response to treatment and any side effects of Therasphere® treatment will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary or metastatic intrahepatic carcinoma
* The cancer must be unresectable with limited established treatment options
* ECOG Performance Status Score 0-2
* Age 19 years or older
* Able to comprehend and provide written informed consent

Exclusion Criteria:

* Any pre-treatment laboratory findings within 15 days of treatment demonstrating:
* Absolute granulocyte count ≤ 1,500/ul
* Platelet count ≤ 75,000/ul
* Serum creatinine > 2.0 mg/dl
* Serum bilirubin ≥ 2.0 mg/dl
* Any of the following contraindications to angiography and selective visceral catheterization:
* History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine
* Bleeding, diathesis, not correctable by usual forms of therapy
* Severe peripheral vascular disease that would preclude catheterization
* Substantial venous shunt away from the liver
* Evidence of potential delivery of greater than 11 mCi (20 Gy absorbed dose) of radiation to the lungs on either 1) first Therasphere® administration; or 2) cumulative delivery of radiation to the lungs over multiple treatments
* Evidence of any detectable Tc-99 MAA flow to the stomach or duodenum, application of established angiographic techniques to stop such flow
* Significant extrahepatic disease representing an imminent life- threatening situation outcome
* Severe liver dysfunction or pulmonary insufficiency
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Pregnant women may not participate

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Russo, MD, Principal Investigator — East Carolina University School of Medicine
Locations (1):
- Leo W Jenkins Cancer Center at East Carolina University School of Medicine, Greenville, North Carolina, United States

REFERENCES:
- [Background] Houle S, Yip TK, Shepherd FA, Rotstein LE, Sniderman KW, Theis E, Cawthorn RH, Richmond-Cox K. Hepatocellular carcinoma: pilot trial of treatment with Y-90 microspheres. Radiology. 1989 Sep;172(3):857-60. doi: 10.1148/radiology.172.3.2549567.
- [Background] Andrews JC, Walker-Andrews SC, Juni JE, Warber S, Ensminger WD. Modulation of liver tumor blood flow with hepatic arterial epinephrine: a SPECT study. Radiology. 1989 Dec;173(3):645-7. doi: 10.1148/radiology.173.3.2813766.
- [Background] Wollner I, Knutsen C, Smith P, Prieskorn D, Chrisp C, Andrews J, Juni J, Warber S, Klevering J, Crudup J, et al. Effects of hepatic arterial yttrium 90 glass microspheres in dogs. Cancer. 1988 Apr 1;61(7):1336-44. doi: 10.1002/1097-0142(19880401)61:73.0.co;2-k. PMID 3345490
- [Background] Ziessman HA, Thrall JH, Gyves JW, Ensminger WD, Niederhuber JE, Tuscan M, Walker S. Quantitative hepatic arterial perfusion scintigraphy and starch microspheres in cancer chemotherapy. J Nucl Med. 1983 Oct;24(10):871-5. PMID 6225839
- [Background] Nakamura H, Tanaka M, Oi H. Hepatic embolization from the common hepatic artery using balloon occlusion technique. AJR Am J Roentgenol. 1985 Jul;145(1):115-6. doi: 10.2214/ajr.145.1.115. No abstract available. PMID 3873830
- [Background] Wellwood JM, Cady B, Oberfield RA. Treatment of primary liver cancer: response to regional chemotherapy. Clin Oncol. 1979 Mar;5(1):25-31. No abstract available. PMID 217565
- [Background] Reed ML, Vaitkevicius VK, Al-Sarraf M, Vaughn CB, Singhakowinta A, Sexon-Porte M, Izbicki R, Baker L, Straatsma GW. The practicality of chronic hepatic artery infusion therapy of primary and metastatic hepatic malignancies: ten-year results of 124 patients in a prospective protocol. Cancer. 1981 Jan 15;47(2):402-9. doi: 10.1002/1097-0142(19810115)47:23.0.co;2-b. PMID 6257376
- [Background] Dusheiko GM, Hobbs KE, Dick R, Burroughs AK. Treatment of small hepatocellular carcinomas. Lancet. 1992 Aug 1;340(8814):285-8. doi: 10.1016/0140-6736(92)92367-o. PMID 1353202
- [Background] Kirk S, Blumgart R, Craig B, Rosen A, Terblanche J, Spence RA. Irresectable hepatoma treated by intrahepatic iodized oil doxorubicin hydrochloride: initial results. Surgery. 1991 Jun;109(6):694-7. PMID 1645890
- [Background] Ravoet C, Bleiberg H, Gerard B. Non-surgical treatment of hepatocarcinoma. J Surg Oncol Suppl. 1993;3:104-11. doi: 10.1002/jso.2930530529. PMID 8389154
- [Background] Audisio RA, Doci R, Mazzaferro V, Bellegotti L, Tommasini M, Montalto F, Marchiano A, Piva A, DeFazio C, Damascelli B, et al. Hepatic arterial embolization with microencapsulated mitomycin C for unresectable hepatocellular carcinoma in cirrhosis. Cancer. 1990 Jul 15;66(2):228-36. doi: 10.1002/1097-0142(19900715)66:23.0.co;2-g. PMID 2164435
- [Background] Ichihara T, Sakamoto K, Mori K, Akagi M. Transcatheter arterial chemoembolization therapy for hepatocellular carcinoma using polylactic acid microspheres containing aclarubicin hydrochloride. Cancer Res. 1989 Aug 1;49(15):4357-62. PMID 2472878
- [Background] Stuart KE, Anand AJ, Jenkins RL. Hepatocellular carcinoma in the United States. Prognostic features, treatment outcome, and survival. Cancer. 1996 Jun 1;77(11):2217-22. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-M. PMID 8635087
- [Background] Di Bisceglie AM, Rustgi VK, Hoofnagle JH, Dusheiko GM, Lotze MT. NIH conference. Hepatocellular carcinoma. Ann Intern Med. 1988 Mar;108(3):390-401. doi: 10.7326/0003-4819-108-3-390. PMID 2449110
- [Background] Kassianides C, Kew MC. The clinical manifestations and natural history of hepatocellular carcinoma. Gastroenterol Clin North Am. 1987 Dec;16(4):553-62. PMID 2831150
- [Background] Gores GJ, Steers JL. Progress in orthotopic liver transplantation for hepatocellular carcinoma. Gastroenterology. 1993 Jan;104(1):317-20. doi: 10.1016/0016-5085(93)90868-d. No abstract available. PMID 8380396
- [Background] Marcos-Alvarez A, Jenkins RL, Washburn WK, Lewis WD, Stuart KE, Gordon FD, Kane RA, Clouse ME. Multimodality treatment of hepatocellular carcinoma in a hepatobiliary specialty center. Arch Surg. 1996 Mar;131(3):292-8. doi: 10.1001/archsurg.1996.01430150070014. PMID 8611095
- [Background] Mazzaferro V, Regalia E, Doci R, Andreola S, Pulvirenti A, Bozzetti F, Montalto F, Ammatuna M, Morabito A, Gennari L. Liver transplantation for the treatment of small hepatocellular carcinomas in patients with cirrhosis. N Engl J Med. 1996 Mar 14;334(11):693-9. doi: 10.1056/NEJM199603143341104. PMID 8594428
- [Background] Selby R, Kadry Z, Carr B, Tzakis A, Madariaga JR, Iwatsuki S. Liver transplantation for hepatocellular carcinoma. World J Surg. 1995 Jan-Feb;19(1):53-8. doi: 10.1007/BF00316980. PMID 7740811
- [Background] Venook AP. Treatment of hepatocellular carcinoma: too many options? J Clin Oncol. 1994 Jun;12(6):1323-34. doi: 10.1200/JCO.1994.12.6.1323. PMID 8201395
- [Background] Ramming KP. The effectiveness of hepatic artery infusion in treatment of primary hepatobiliary tumors. Semin Oncol. 1983 Jun;10(2):199-205. No abstract available. PMID 6306834
- [Background] Nerenstone S, Friedman M. Medical treatment of hepatocellular carcinoma. Gastroenterol Clin North Am. 1987 Dec;16(4):603-12. PMID 2831153
- [Background] Solomon B, Soulen MC, Baum RA, Haskal ZJ, Shlansky-Goldberg RD, Cope C. Chemoembolization of hepatocellular carcinoma with cisplatin, doxorubicin, mitomycin-C, ethiodol, and polyvinyl alcohol: prospective evaluation of response and survival in a U.S. population. J Vasc Interv Radiol. 1999 Jun;10(6):793-8. doi: 10.1016/s1051-0443(99)70117-x. PMID 10392950
- [Background] BREEDIS C, YOUNG G. The blood supply of neoplasms in the liver. Am J Pathol. 1954 Sep-Oct;30(5):969-77. No abstract available. PMID 13197542
- [Background] SCHENK WG Jr, McDONALD JC, McDONALD K, DRAPANAS T. Direct measurement of hepatic blood flow in surgical patients: with related observations on hepatic flow dynamics in experimental animals. Ann Surg. 1962 Sep;156(3):463-71. doi: 10.1097/00000658-196209000-00013. No abstract available. PMID 14498225
- [Background] Sasaki Y, Imaoka S, Kasugai H, Fujita M, Kawamoto S, Ishiguro S, Kojima J, Ishikawa O, Ohigashi H, Furukawa H, et al. A new approach to chemoembolization therapy for hepatoma using ethiodized oil, cisplatin, and gelatin sponge. Cancer. 1987 Sep 15;60(6):1194-203. doi: 10.1002/1097-0142(19870915)60:63.0.co;2-t. PMID 2441837
- [Background] Yamada R, Kishi K, Sato M, Sonomura T, Nishida N, Tanaka K, Shioyama Y, Terada M, Kimura M. Transcatheter arterial chemoembolization (TACE) in the treatment of unresectable liver cancer. World J Surg. 1995 Nov-Dec;19(6):795-800. doi: 10.1007/BF00299773. PMID 8553668
- [Background] Madden MV, Krige JE, Bailey S, Beningfield SJ, Geddes C, Werner ID, Terblanche J. Randomised trial of targeted chemotherapy with lipiodol and 5-epidoxorubicin compared with symptomatic treatment for hepatoma. Gut. 1993 Nov;34(11):1598-600. doi: 10.1136/gut.34.11.1598. PMID 8244149
- [Background] Groupe d'Etude et de Traitement du Carcinome Hepatocellulaire. A comparison of lipiodol chemoembolization and conservative treatment for unresectable hepatocellular carcinoma. N Engl J Med. 1995 May 11;332(19):1256-61. doi: 10.1056/NEJM199505113321903. PMID 7708069
- [Background] Pelletier G, Roche A, Ink O, Anciaux ML, Derhy S, Rougier P, Lenoir C, Attali P, Etienne JP. A randomized trial of hepatic arterial chemoembolization in patients with unresectable hepatocellular carcinoma. J Hepatol. 1990 Sep;11(2):181-4. doi: 10.1016/0168-8278(90)90110-d. PMID 2174933
- [Background] Bruix J, Llovet JM, Castells A, Montana X, Bru C, Ayuso MC, Vilana R, Rodes J. Transarterial embolization versus symptomatic treatment in patients with advanced hepatocellular carcinoma: results of a randomized, controlled trial in a single institution. Hepatology. 1998 Jun;27(6):1578-83. doi: 10.1002/hep.510270617. PMID 9620330
- [Background] Uchida M, Kohno H, Kubota H, Hayashi T, Yamanoi A, Kimoto T, Ono T, Nagasue N. Role of preoperative transcatheter arterial oily chemoembolization for resectable hepatocellular carcinoma. World J Surg. 1996 Mar-Apr;20(3):326-31. doi: 10.1007/s002689900052. PMID 8661839
- [Background] Stuart K, Stokes K, Jenkins R, Trey C, Clouse M. Treatment of hepatocellular carcinoma using doxorubicin/ethiodized oil/gelatin powder chemoembolization. Cancer. 1993 Dec 1;72(11):3202-9. doi: 10.1002/1097-0142(19931201)72:113.0.co;2-4. PMID 7694787
- [Background] Berger DH, Carrasco CH, Hohn DC, Curley SA. Hepatic artery chemoembolization or embolization for primary and metastatic liver tumors: post-treatment management and complications. J Surg Oncol. 1995 Oct;60(2):116-21. doi: 10.1002/jso.2930600210. PMID 7564377
- [Background] Vetter D, Wenger JJ, Bergier JM, Doffoel M, Bockel R. Transcatheter oily chemoembolization in the management of advanced hepatocellular carcinoma in cirrhosis: results of a Western comparative study in 60 patients. Hepatology. 1991 Mar;13(3):427-33. PMID 1847892
- [Background] Perry LJ, Stuart K, Stokes KR, Clouse ME. Hepatic arterial chemoembolization for metastatic neuroendocrine tumors. Surgery. 1994 Dec;116(6):1111-6; discussion 1116-7. PMID 7985095
- [Background] Ehrhardt GJ, Day DE. Therapeutic use of 90Y microspheres. Int J Rad Appl Instrum B. 1987;14(3):233-42. doi: 10.1016/0883-2897(87)90047-x. PMID 3667306
- [Background] Mantravadi RV, Spigos DG, Tan WS, Felix EL. Intraarterial yttrium 90 in the treatment of hepatic malignancy. Radiology. 1982 Mar;142(3):783-6. doi: 10.1148/radiology.142.3.7063703. No abstract available.
- [Background] Herba MJ, Illescas FF, Thirlwell MP, Boos GJ, Rosenthall L, Atri M, Bret PM. Hepatic malignancies: improved treatment with intraarterial Y-90. Radiology. 1988 Nov;169(2):311-4. doi: 10.1148/radiology.169.2.3174978.
- [Background] Blanchard RJ, Morrow IM, Sutherland JB. Treatment of liver tumors with yttrium-90 microspheres alone. Can Assoc Radiol J. 1989 Aug;40(4):206-10. PMID 2766018
- [Background] Andrews JC, Walker SC, Ackermann RJ, Cotton LA, Ensminger WD, Shapiro B. Hepatic radioembolization with yttrium-90 containing glass microspheres: preliminary results and clinical follow-up. J Nucl Med. 1994 Oct;35(10):1637-44. PMID 7931662
- [Background] BLANCHARD RJ, GROTENHUIS I, LAFAVE JW, PERRY JF Jr. BLOOD SUPPLY TO HEPATIC V2 CARCINOMA IMPLANTS AS MEASURED BY RADIOACTIVE MICROSPHERES. Proc Soc Exp Biol Med. 1965 Feb;118:465-8. doi: 10.3181/00379727-118-29876. No abstract available. PMID 14268654
- [Background] Stribley KV, Gray BN, Chmiel RL, Heggie JC, Bennett RC. Internal radiotherapy for hepatic metastases II: The blood supply to hepatic metastases. J Surg Res. 1983 Jan;34(1):25-32. doi: 10.1016/0022-4804(83)90018-5. PMID 6681644
- [Background] Gyves JW, Ziessman HA, Ensminger WD, Thrall JH, Niederhuber JE, Keyes JW Jr, Walker S. Definition of hepatic tumor microcirculation by single photon emission computerized tomography (SPECT). J Nucl Med. 1984 Sep;25(9):972-7. PMID 6088735
- [Background] Chamberlain MN, Gray BN, Heggie JC, Chmiel RL, Bennett RC. Hepatic metastases--a physiological approach to treatment. Br J Surg. 1983 Oct;70(10):596-8. doi: 10.1002/bjs.1800701009. PMID 6626920
- [Background] Meade VM, Burton MA, Gray BN, Self GW. Distribution of different sized microspheres in experimental hepatic tumours. Eur J Cancer Clin Oncol. 1987 Jan;23(1):37-41. doi: 10.1016/0277-5379(87)90416-0. PMID 3595684
- [Background] Chuang VP. Hepatic tumor angiography: a subject review. Radiology. 1983 Sep;148(3):633-9. doi: 10.1148/radiology.148.3.6878677.
- [Background] Leung TW, Lau WY, Ho SK, Ward SC, Chow JH, Chan MS, Metreweli C, Johnson PJ, Li AK. Radiation pneumonitis after selective internal radiation treatment with intraarterial 90yttrium-microspheres for inoperable hepatic tumors. Int J Radiat Oncol Biol Phys. 1995 Nov 1;33(4):919-24. doi: 10.1016/0360-3016(95)00039-3. PMID 7591903
- [Background] YA PM, GUZMAN T, LOKEN MK, PERRY JF Jr. Isotope localization with tagged microspheres. Surgery. 1961 May;49:644-50. No abstract available. PMID 13787028
- [Background] LAFAVE JW, GROTENHUIS I, KIM YS, MACLEAN LD, PERRY JF Jr. Y90-tagged microspheres in adjuvant tumor therapy. Surgery. 1963 Jun;53:778-83. No abstract available. PMID 13928002
- [Background] GRADY ED, SALE WT, ROLLINS LC. Localization of radioactivity by intravascular injection of large radioactive particles. Ann Surg. 1963 Jan;157(1):97-114. doi: 10.1097/00000658-196301000-00012. No abstract available. PMID 13949718
- [Background] BLANCHARD RJ, GROTENHUIS I, LAFAVE JW, FRYE CW, PERRY JF Jr. TREATMENT OF EXPERIMENTAL TUMORS; UTILIZATION OF RADIOACTIVE MICROSPHERES. Arch Surg. 1964 Aug;89:406-10. doi: 10.1001/archsurg.1964.01320020170025. No abstract available. PMID 14160169
- [Background] Stribley KV, Gray BN, Chmiel RL, Heggie JC, Bennett RC. Internal radiotherapy for hepatic metastases I: The homogeneity of hepatic arterial blood flow. J Surg Res. 1983 Jan;34(1):17-24. doi: 10.1016/0022-4804(83)90017-3. PMID 6823100
- [Background] Mauderly JL, Pickrell JA, Hobbs CH, Benjamin SA, Hahn FF, Jones RK, Barnes JE. The effects of inhaled 90Y fused clay aerosol on pulmonary function and related parameters of the beagle dog. Radiat Res. 1973 Oct;56(1):83-96. No abstract available. PMID 4743733
- [Background] Hill JW, Whitehead WS, Cameron JD, Hedgecock GA. Glass fibres: absence of pulmonary hazard in production workers. Br J Ind Med. 1973 Apr;30(2):174-9. doi: 10.1136/oem.30.2.174. PMID 4703089
- [Background] Russell JL Jr, Carden JL, Herron HL. Dosimetry calculations for yttrium-90 used in the treatment of liver cancer. Endocurietherapy/Hyperthermia Oncology. 1988; 4:171-186.
- [Background] Boos G, Thirwell M, Blanchard R, et al. Phase I-II study of hepatic arterial infusion of yttrium-90 (Y-90) glass microspheres in cancer of the liver. Proc Am Soc Clin Oncol. 1989, 8:103.
- [Background] Patt YZ, Charnsangavej C, Boddie A, et al. Treatment of hepatocellular carcinoma with hepatic arterial floxuridine, doxorubicin, and mitomycin C (FUDRM) with or without hepatic arterial embolization: factors associated with longer arterial survival. Reg Cancer Treat. 1989; 2:98.
- [Background] Douglass C. Prolongation of survival with periodic percutaneous multi-drug arterial infusions in patients with primary and metastatic gastrointestinal carcinoma to liver, abstracted. Proc Am Soc Clin Oncol. 1980; 21:416
- [Background] Stuart K. Invited commentary on preoperative lipiodol for unresectable HCC. World J Surg 1996; 20:331
- [Background] Harbert JC, Ziessman HA. Therapy with intra-arterial microspheres. Nuclear Medicine Annual 1987, edited by Freeman L.M., Weissman H.S. Raven Press, New York.
- [Background] Dancey JE, Shepherd FA, Paul K, Sniderman KW, Houle S, Gabrys J, Hendler AL, Goin JE. Treatment of nonresectable hepatocellular carcinoma with intrahepatic 90Y-microspheres. J Nucl Med. 2000 Oct;41(10):1673-81. PMID 11037997
- [Background] PRINZMETAL M, SIMKIN B, et al. Studies on the coronary circulation; the collateral circulation of the normal human heart by coronary perfusion with radioactive erythrocytes and glass spheres. Am Heart J. 1947 Apr;33(4):420-42. doi: 10.1016/0002-8703(47)90090-2. No abstract available. PMID 20292386
- [Background] Prinzmetal M, Ornitz EM Jr. Arterio-venous anastomoses in liver, spleen, and lungs. Am J Physiol. 1948 Jan 1;152(1):48-52. doi: 10.1152/ajplegacy.1947.152.1.48. No abstract available. PMID 18903426
- [Background] Gross P. The effects of fibrous glass dust on the lungs of animals. In: Occupational exposure to fibrous glass of a symposium presented to the Center of Adult Education; 1976; University of Maryland, College Park, MD. 169-178.